CLINICAL TRIAL: NCT01156506
Title: Patient Perspectives on Living With an Enterostoma and Rehabilitation
Brief Title: Focus Group Interviews of Patients With Permanent or Temporary Enterostomas
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Anne Kjærgaard Danielsen, Ph.d.student, RN, Herlev Hospital
Other Study IDs: AKD02
Record Dates: First submitted 2010-06-30; First posted 2010-07-05 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Patient Perspective; Living With an Enterostoma; Mastery; Empowerment
Keywords: quality of life; patient education; rehabilitation; focus group interview
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The study seeks to gain knowledge about new and of alternative ways of organizing ostomy training based on informants' own experiences of life with a stoma.

The study is designed and conducted as qualitative focus group interviews with three different groups of patients with enterostomas (5-8 in each group): a) people with permanent enterostoma due to cancer, 2) people with permanent enterostoma due to non-cancer and 3) people with a temporary ileostomy.

DETAILED DESCRIPTION:
The study is investigating the perspective of the patients who have actually experienced having surgery and living with an enterostoma.

By applying this method it is possible to gain access and in depth knowledge of complex issues including sensitive data. The dialogue with peers can lead to experiments and associations which might stimulate the informants to produce new insights within the individual and in the group.

The interviews will be transcribed in full and analyzed with qualitative content analysis with a phenomenological and hermeneutical approach

ELIGIBILITY:
Inclusion Criteria:

* Patients with permanent enterostoma due to cancer.
* Patients with permanent enterostoma due to other causes.
* Patients with temporary ileostomy.

Exclusion Criteria:

* Patients with severe mental disorders.
* Patients who do not communicate in Danish.
* Patients with severe hearing impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of surgery
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Educational elements and themes that will optimize rehabilitation and patient education | up until 10 months from interview
  Illumination and discussion of informants´ perspective on rehabilitation and patient education will

SECONDARY OUTCOMES:
Identification of strategies for improving quality of life | up until 10 months from interview
  Illumination and discussion of informants perspective on the influence of an enterostoma on their lives

CONTACTS AND LOCATIONS:
Overall Officials: Anne K. Danielsen, Nurse, MaClN, Principal Investigator — Herlev University Hospital, department of surgery